CLINICAL TRIAL: NCT02823639
Title: Efficacy and Mechanisms of Transcranial Direct Current Stimulation (tDCS) - Effects on Working Memory in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Munich (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Prof. Dr., University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 01EE1407H
Record Dates: First submitted 2016-06-20; First posted 2016-07-06 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anodal Stimulation tDCS; Schizophrenia; Working Memory
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial direct current stimulation (Active Comparator): tDCS with varying intensity, location and polarity
  Interventions: Procedure: Transcranial direct current stimulation
- Sham stimulation (Placebo Comparator): Double blind sham stimulation with sham mode of neuroConn device
  Interventions: Procedure: Transcranial direct current stimulation

INTERVENTIONS:
Procedure: Transcranial direct current stimulation
  Other Names: tDCS

SUMMARY:
Impairments of cognition are a core, severely disabling feature of schizophrenia leading to poor long-term outcome with no established treatment available.

Particularly impaired executive functions (e.g working memory) are frequently observed and are consistently associated with reduced activation of the dorsolateral prefrontal cortex (dlPFC). Deficits in those functions have been shown to be closely related to negative symptoms, thought disorder, and functional outcome in schizophrenia leading to the notion that frontal lobe dysfunction is crucially important in schizophrenic psychopathology.

Noninvasive brain stimulation like tDCS can enhance executive functions like working memory in healthy subjects as well as in patients. To identify the optimal parameters for this intervention in patients with schizophrenia, the investigators first test the effects of different polarities (anodal, cathodal), stimulation intensities (1mA, 2mA) and laterality (left, right) on working-memory performance (nback task) in a sham-controlled cross-over design (n=128). To elucidate mechanisms of action, oscillatory brain activity will be registered with electroencephalography (EEG).

These experiments will provide reliable data for an evidence-based development of new clinical interventions to improve treatment of cognitive deficits in patients with schizophrenia and thus enhance schizophrenia prevention and recovery.

DETAILED DESCRIPTION:
1. Working hypothesis:

   In patients with subacute schizophrenia, transcranial direct current stimulation (tDCS) to the dorsolateral prefrontal cortex (dlPFC) exerts lasting beneficial effects on working-memory performance.
2. Research question(s):

   In patients with remitted early phase schizophrenia, this research project aims at providing evidence for:

   i) immediate improvement of working-memory performance by application of tDCS to the dlPFC in patients with schizophrenia; ii) determination of the optimal stimulation polarity, dosage and localization; iii) neurophysiological mechanisms (modulation in oscillatory activity and functional connectivity) and predictors of tDCS effects; iv) modulating effect of gender on the malleability of executive functions with tDCS.
3. Previous work of the investigators:

   The investigators have provided proof-of principle evidence for persisting improvement of cognitive planning by a polarity-specific learning-stage dependent coupling of training and stimulation. The investigators have demonstrated that working memory and deficient cognitive control can be enhanced with anodal tDCS in depression and that the effects of tDCS are modulated by genetic polymorphisms. The investigators were the first to show impaired cortical plasticity following tDCS in schizophrenia patients at different disease states. Finally, the investigators have just successfully finished the world-wide largest clinical trial investigating the efficacy of non-invasive brain stimulation (rTMS) on negative symptoms in schizophrenia (DFG 241/10-1, Falkai, Hasan).
4. Aims and work plan:

To examine the potential of tDCS for the improvement of working memory with remitted schizophrenia the investigators are following this work plan:

I) Immediate effects on performance:

Assessment of efficacy of tDCS polarity (anodal, cathodal), dosage (1mA, 2mA) and laterality (left and right dlPFC) on working memory (adaptive n-back(6)) in patients (n=2x2x2x16=128). In a two-session cross-over design, stimulation (tDCS and sham) will be applied to the dlPFC (left or right) for 20min (during task performance).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed schizophrenia (DSM-V)
* age (18 - 60 years)
* right handedness
* stable medication during 1 week of treatment and 1 week before

Exclusion Criteria:

* history of seizures
* metal device throughout the body
* pregnancy
* use of anticonvulsive medication
* use of benzodiazepines more than 1 mg of Lorazepam equivalent
* current substance abuse (nicotine excluded)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-10; Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change of dprime | Assessment during stimulation in a n-back task at three specific timepoints during one week
  dprime provides the separation between the means of the signal and the noise distributions, compared against the standard deviation of the signal plus noise distributions

SECONDARY OUTCOMES:
Change of reaction time in n-back task | Assessment during stimulation in a n-back task at three specific timepoints during one week

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, Prof., MD, Principal Investigator — University Hospital Tuebingen, Department of Psychiatry and Psychotherapy
Locations (2):
- Germany (2):
  - LMU Muenchen, Department of Psychiatry and Psychotherapy, München
  - University Hospital Tuebigen, Department of Psychiatry and Psychotherapy, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided